CLINICAL TRIAL: NCT00003367
Title: The Effect of a Low Fat Diet, High in Soy, Fruits, Vegetables, Green Tea, Vitamin E and Fiber on the PSA in Patients With Prostate Cancer
Brief Title: Diet and PSA Levels in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 98-014; CDR0000066354 (Registry Identifier: PDQ (Physician Data Query)); NCI-G98-1445
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Tea; Soybean Proteins; Vitamin E

INTERVENTIONS:
Dietary Supplement: green tea
Dietary Supplement: soy protein isolate
Dietary Supplement: vitamin E

SUMMARY:
RATIONALE: The amount of fat, fiber, soy, fruits, vegetables, vitamin E, and green tea in the diet may affect androgen metabolism in men. This may affect PSA level in patients with prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two diets, differing in fat, fiber, soy, fruit, vegetable, vitamin E, and green tea content, in affecting PSA level in patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effects of 2 dietary regimens on levels of prostate-specific antigen (PSA) in patients with prostate cancer. II. Determine the compliance of these patients with the dietary regimen. III. Evaluate the effects of the dietary regimen on quality of life in these patients. IV. Evaluate the effects of the dietary regimen on PSA anxiety in these patients. V. Evaluate the effects of the dietary regimen on obesity, high blood pressure, and serum cholesterol in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to previous treatment (prostatectomy vs radiotherapy) and prostate-specific antigen (PSA) level (less than 5 mg/mL vs 5 or greater mg/mL). All patients complete quality of life, dietary, and other questionnaires before, during, and at the conclusion of the study. Patients are randomized to one of two dietary intervention regimens: Arm I (Intensive Nutritional Intervention): Patients are assigned to follow a low fat, high fiber diet that is also high in soy, fruits and vegetables, green tea, and vitamin E. Patients meet with a nutritionist for nutrition education and dietary counseling weekly for 8 weeks, then every 2 weeks for 2 months, and then monthly for 14 months. Sessions include dietary counseling, meal planning, and instruction in skills necessary to maintain dietary lifestyle changes. Patients record their dietary intake on a regular basis. Arm II (General Nutritional Instruction): Patients are assigned to follow dietary guidelines established by the National Cancer Institute. Patients meet with a nutritionist for dietary counseling and monitoring every 2 months for 18 months. Patients on both arms have PSA levels tested before the study, 1 and 3 months into the study, and then every 3 months thereafter for up to 18 months.

PROJECTED ACCRUAL: A total of 154 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate with either: Two increases in prostate-specific antigen (PSA) levels with a minimal 30% increase in range of values following either prostate surgery (prostatectomy) or radiation therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: At least 6 months Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 2.0 mg/dL OR SGOT less than 3 times upper limit of normal (ULN) Renal: Creatinine less than 2.0 mg/dL OR Creatinine clearance greater than 40 mL/min Cardiovascular: No significant heart disease (New York Heart Association class III or IV) Pulmonary: No severe debilitating pulmonary disease Other: No narcotic dependent pain No extreme dietary patterns (such as a macrobiotic diet) No baseline diet having fewer than 25% calories from fat No history of second malignancy within past 5 years except nonmelanomatous skin cancer No insulin-dependent diabetes No infection requiring antibiotics

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: At least 4 weeks since hormone therapy Radiotherapy: At least 4 weeks since radiotherapy Surgery: Prior prostatectomy allowed Other: Recovered from toxic effects of any prior therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 1998-04; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Shike, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States